CLINICAL TRIAL: NCT01694719
Title: Cognitive Control Training as an Adjunct to Behavioral Activation Therapy in the Treatment of Depression
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Boston University (Other)
Responsible Party: Principal Investigator, Samantha Moshier, M.A., Doctoral Candidate in Psychology, Boston University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2930
Record Dates: First submitted 2012-09-24; First posted 2012-09-27 (Estimated); Last update posted 2012-09-27 (Estimated); Status verified 2012-09

CONDITIONS: Depression
Keywords: Depression; Major Depressive Disorder; Behavioral Activation; Cognitive Training
MeSH Terms: conditions — Depression; Depressive Disorder, Major

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Behavioral Activation + Cognitive Control Training (Experimental): Participants will receive 5 sessions of behavioral activation therapy concurrent with 4 sessions of cognitive control training, a computerized intervention which targets cognitive control processes such as working memory and attention.
  Interventions: Behavioral: Brief Behavioral Activation Treatment for Depression; Behavioral: Cognitive Control Training
- Behavioral Activation Therapy plus Control Task (Active Comparator): Participants will receive 5 sessions of behavioral activation therapy and 4 sessions of a non-active, computerized control task.
  Interventions: Behavioral: Brief Behavioral Activation Treatment for Depression

INTERVENTIONS:
Behavioral: Brief Behavioral Activation Treatment for Depression
Behavioral: Cognitive Control Training
  Arms: Behavioral Activation + Cognitive Control Training

SUMMARY:
The purpose of this study is to evaluate the potential effects of a cognitive training program when combined with a particular form of psychotherapy (behavioral activation therapy) for depression. Behavioral activation therapy targets changes in behavior as a method for improving a depressed individual's thoughts, feelings, and overall quality of life. This study is designed to test whether a computerized brain exercise called cognitive control training can enhance the effects of a 5-session behavioral activation therapy program. CCT has been shown to reduce depressive symptoms in two other studies, but it has not yet been combined with behavioral activation therapy. The investigators hypothesize that individuals assigned to the behavioral activation plus cognitive control training condition will demonstrate reduced depressive symptoms from pre to post treatment compared with those assigned to the behavioral activation plus computerized control condition. The investigators hypothesize that these gains will be maintained at one-month follow up.

ELIGIBILITY:
Inclusion Criteria:

1. Adults ages 18-65
2. Primary psychiatric diagnosis of major depressive disorder
3. Ability to read and speak English sufficiently to complete study procedures
4. If taking antidepressant or anxiolytic medication, participants must be taking a stabilized dose for a minimum period of at least 8 weeks prior to entry into the study
5. Willingness and ability to comply with the requirements of the study protocol

Exclusion Criteria:

1. Lifetime history of bipolar disorder or psychotic disorder
2. Neurological disorder such as Parkinson's disease or traumatic brain injury
3. Alcohol or substance dependence within the past 6 months
4. Substantial suicide risk
5. Concurrent psychotherapy initiated within 2 months of baseline, or ongoing psychotherapy of any duration directed specifically toward treatment of the depression other than general supportive therapy
6. Current use of antipsychotics, stimulants, or modafinil

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Estimated)
Dates: Start 2012-09; Primary Completion 2013-10 (Estimated); Study Completion 2013-10 (Estimated)

PRIMARY OUTCOMES:
Beck Depression Inventory

SECONDARY OUTCOMES:
Montgomery Asberg Depression Rating Scale

OTHER OUTCOMES:
Ruminative Response Scale

CONTACTS AND LOCATIONS:
Locations (1):
- Boston University - Translational Research Program, Boston, Massachusetts, United States